CLINICAL TRIAL: NCT01550900
Title: A Prospective Placebo-control Double-blind Randomized Trial of Metformin in Chemoprevention of Metachronous Colonic Neoplastic Polyps
Brief Title: Prospective Trial of Metformin - Chemoprevention Role
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-1100
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Colorectum
Keywords: Colorectum; Metachronous ctalColonic Neoplastic Polyps; Chemoprevention; Colonic adenoma(s); Pre-cancerous tumor(s) on the colon; Metformin ER; Extended Release; Placebo; Sugar pill
MeSH Terms: interventions — Metformin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin ER (Experimental): Participants receive two tablets of Metformin ER 500 mg once daily for no more than twelve to eighteen months allowing time for at least one follow up colonoscopy. Dose will be reached in a gradual escalation scheme to improve gastrointestinal tolerance. If participants experience side effects during dose escalation regimen, they will be reduced to one tablet of 500 mg daily, and may continue taking 500 mg daily for the duration of the study.
  Interventions: Drug: Metformin ER
- Placebo (Active Comparator): Control group given matched Placebo once daily for no more than twelve to eighteen months allowing time for at least one follow up colonoscopy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin ER — Starting dose: 500 mg by mouth daily for 1 week with weekly increases of 250 mg daily to target dose of 1000 mg daily.
  Arms: Metformin ER
Other: Placebo — Placebo tablets by mouth 1 time a day.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The goal of this clinical research study is to learn if metformin extended release (ER) can prevent colonic adenomas from becoming cancerous. Metformin ER will be compared to a placebo.

Metformin ER is designed to block a protein in tumor cells that is important in tumor growth and blood vessel development. This may cause cell death or reduce the spread of the disease.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Colonic adenomas are considered pre-cancerous, but they may change into colorectal cancer. Patients have a higher risk of developing additional adenomas if adenomas are found at the time of their follow-up colonoscopy.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being assigned to either group.

If you are in Group 1, you will receive metformin ER

If you are in Group 2, you will receive a placebo.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You will take metformin ER/placebo tablets by mouth 1 time a day with food for 12-18 months (usually 12 months but sometimes up to 18 if the doctor thinks it is needed). This will allow time for at least 1 repeat follow-up colonoscopy.

The dose of metformin ER will be increased at Week 2 and again at Week 3. If you have side effects, the dose may be lowered if the doctor thinks it is needed.

Study Visit:

At 3-12 months or 3-18 months after you start taking metformin ER/placebo, you will have another colonoscopy and standard tissue collection for colonic adenoma(s). This tissue will be used for biomarker testing. Blood (about 3 tablespoons) will be drawn for testing on your blood sugar and for biomarker testing. You will need to fast for 8 hours before this test.

Your blood and tissue will also be used for research on the cause of colorectal cancer and biomarker testing.

Length of Treatment:

You may continue taking the study drug for 12 months. However, if your doctor thinks it is needed, a follow-up colonoscopy may be scheduled for you at either 15 or 18 months after enrollment. If this is the case, you will continue taking the drug for up to 18 months. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the study visit.

This is an investigational study. Metformin ER is FDA approved and commercially available for the treatment of type 2 diabetes. Its use to prevent colonic adenomas is investigational.

Up to 128 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 75 years
2. Polyp features suggesting high risk for recurrence include: piece-meal polypectomy, large (>10mm) neoplastic polyp, polyp with high grade dysplasia, or substantial number (>10) of neoplastic polyps.
3. ability to give informed consent
4. Patients should be registered on LAB10-0417
5. Diabetic patients are eligible but they may be excluded if they are taken Metformin, insulin or sulfonylureas

Exclusion Criteria:

1. Patients with renal insufficiency defined as serum creatinine >= 1.4 mg/dl for females and >= 1.5 mg/dl for males by the manufacturer.
2. Pregnant or nursing women
3. A malignancy currently under active therapy
4. Unstable angina, uncontrolled ischemic cardiac disease or symptomatic congestive heart failure (e.g. Class III or IV New York Heart Association's Functional Classification)
5. Current usage of Metformin
6. Current usage of insulin, sulfonylureas
7. History of lactic acidosis
8. Liver dysfunction including chronic active hepatitis and cirrhosis
9. Inability to give informed consent
10. Other investigational drugs within the past one year or concurrently
11. Known hypersensitivity or intolerance to Metformin
12. Contraindications for repeat colonoscopy
13. Inflammatory bowel disease
14. Rectosigmoiditis of any etiology

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Ki-67-Stained Nuclei in Normal Rectal Mucosa | 3 months
  Primary endpoint defined as change in overall proliferation index between baseline and first return visit, that is, percentage of Ki-67-stained nuclei, in normal rectal mucosa. Tissue samples will be obtained at baseline colonoscopy and subsequent exams for analysis including Ki67, caspase 3, and various biomarkers and immunohistochemicals studies.

CONTACTS AND LOCATIONS:
Overall Officials: William Ross, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org